CLINICAL TRIAL: NCT00761813
Title: Fixation Using Alternative Implants for the Treatment of Hip Fractures: A Multi-Centre Randomized Trial Comparing Sliding Hip Screws and Cancellous Screws on Revision Surgery Rates and Quality of Life in the Treatment of Femoral Neck Fractures
Brief Title: Using Alternative Implants for the Surgical Treatment of Hip Fractures (The FAITH Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Stichting Nuts Ohra (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR055267 (NIH); R01AR055267 (NIH); NCT00557167 (obsolete NCT alias)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Femoral Neck Fractures
Keywords: Sliding Hip Screw Fixation; Cannulated Screw Fixation
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Sliding Hip Screw (Experimental)
  Interventions: Device: Open reduction internal fixation (ORIF) with single sliding hip screw
- Multiple Cancellous Screws (Experimental)
  Interventions: Device: ORIF with multiple cancellous screws

INTERVENTIONS:
Device: Open reduction internal fixation (ORIF) with single sliding hip screw — The ORIF will be performed using a single large diameter partially threaded screw that is affixed to the proximal femur with a side plate (with a minimum of two holes and a maximum of four holes) and no supplemental fixations. Surgeons will use any commercially available sliding hip screw implant and will insert implants as per the manufacturers' technical guides. Other surgical factors will be based on surgeon preference and noted.
  Arms: Single Sliding Hip Screw
Device: ORIF with multiple cancellous screws — ORIF will be performed using multiple small diameter threaded screws (with a minimum of two screws and a minimum diameter of 6.5 mm). Surgeons will use any threaded screw or hook pin and will follow the manufacturers' technical guides. Other surgical factors will be based on surgeon preference and noted.
  Arms: Multiple Cancellous Screws

SUMMARY:
Each year, hip fracture, an injury that can impair independence and quality of life, occurs in about 280,000 Americans and 36,000 Canadians. The annual healthcare costs associated with this injury are expected to soon reach $9.8 billion in the United States and $650 million in Canada. It is important to have in place optimal practice guidelines for the surgical handling of this injury. One type of hip fracture, called a femoral neck fracture, is often treated with a surgical procedure called internal fixation. When performing internal fixation, most orthopaedic surgeons favor using multiple small diameter screws over using a single large diameter screw with a sliding plate. However, use of the sliding hip screw might in fact result in fewer complications after surgery and reduce the need for a second surgery, called a revision surgery. This study will compare the two different surgical procedures to determine which one results in better outcomes after surgery.

DETAILED DESCRIPTION:
One type of hip fracture, called a femoral neck fracture, involves a break in the narrow part of the femur bone where the head of the femur is joined to the main shaft. The break can be either undisplaced, which involves very little separation at the fracture site, or displaced, in which there is substantial separation. Surgeons agree that the best surgical procedure for an undisplaced fracture is internal fixation, in which a mechanical implant reconnects the two separated segments of bone. For displaced fractures, surgeons usually choose between internal fixation and a hip joint replacement.

There is more than one way to perform internal fixation. The majority of orthopaedic surgeons currently favor the use of multiple small diameter cancellous screws. However, an alternative method that uses a single large diameter screw attached to a sideplate, called a sliding hip screw, has been gaining popularity and might reduce post-surgical complications and the need for revision surgery. Which surgical method is best for the patient is unknown. This study will compare the use of multiple small diameter cancellous screws versus a single sliding hip screw on rates of revision surgery 2 years after patients sustain femoral neck fractures and undergo internal fixation. The study will also compare the impact of the two different surgical procedures on the overall health, function, and quality of life of patients. Results from this study may impact current orthopaedic practice.

Participation in this study will last 2 years. Before surgery, participants will complete a baseline assessment that will include x-rays, a medical history review, and a physical examination. Participants will then be randomly assigned to undergo one of two types of internal fixation surgeries for repairing their hip fractures. In one group of participants, surgeons will use at least two small cancellous threaded screws that have a diameter of at least 6.5 mm. In the other group of participants, surgeons will use a single large diameter screw that is partially threaded. This screw, called a sliding hip screw, will be affixed to the femur bone with a sideplate, and there will be no other fixations. All surgeons, who will need to meet certain criteria to partake in the study, will follow the manufacturers' technique guidelines for using either type of screw. Specific aspects of both the pre-operative and post-operative care, such as the use of antibiotics and calcium supplementation, will be standardized for all participants.

Follow-up assessments will be completed either by phone or in-person at the hospital or clinic. They will occur 1, 2, and 10 weeks after surgery and 6, 9, 12, 18, and 24 months after surgery. All assessments will include questionnaires and interviews on health status, hip function, pain, and revision surgery. Some of the in-person assessments will also include x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of femoral neck
* Operative treatment within 4 days for displaced fractures
* Operative treatment within 7 days for nondisplaced fractures
* Ambulatory before the injury
* Low energy trauma, such as falls from a sitting or standing position
* No other major trauma

Exclusion Criteria:

* Unsuited for both surgical treatments
* Associated major injuries of the lower extremities
* Retained hardware around the hip
* Infection around the hip
* Bone metabolic disorder (except for osteoporosis)
* Moderate or severe cognitive impairment
* Parkinson's disease or dementia
* Unable to complete the 2-year follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2009-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Swiontkowski, MD, Principal Investigator — University of Minnesota; Mohit Bhandari, MD, Principal Investigator — McMaster University
Locations (32):
- United States (32):
  - University of Alabama @ Birmingham, Birmingham, Alabama
  - Kamran Aurang, MD, Irvine, California
  - University of Califnornia-Irvine, Orange, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Mark Hammerberg, Denver, Colorado
  - Rocky Mountain Orthopaedic/Western Slope Study Group, Grand Junction, Colorado
  - Indiana University-Wishard Hlth Serv., Indianapolis, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Orthopaedic Associates of Grand Rapids, Grand Rapids, Michigan
  - Colleen Linehan, MD, Saginaw, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota-Regions Hospital, Saint Paul, Minnesota
  - Columbia Orthopaedic Group, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - Robert Wood Johnson University, New Brunswick, New Jersey
  - University of Rochester Med. Ctr., Rochester, New York
  - Mission Hospital Res. Unit, Asheville, North Carolina
  - Univ. of Cincinnati Med Ctr, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Humility of Mary Health Partners/St. Elizabeth Hlth Ctr, Youngstown, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Vanderbilt University Orthopaedic Instititute, Nashville, Tennessee
  - US Army Institute of Surgical Research, Fort Sam Houston, Texas
  - Texas Tech Univ. Hlth Sci. Ctr., Lubbock, Texas
  - University of Texas HSC (San Antonio), San Antonio, Texas
  - Scott & White Hospital, Temple, Texas
  - Northwest Orthopaedic Specialists, Spokane, Washington

REFERENCES:
- [Derived] van de Kuit A, Oosterhoff JHF, Dijkstra H, Sprague S, Bzovsky S, Bhandari M, Swiontkowski M, Schemitsch EH, IJpma FFA, Poolman RW, Doornberg JN, Hendrickx LAM; , the Machine Learning Consortium and FAITH Investigators. Patients With Femoral Neck Fractures Are at Risk for Conversion to Arthroplasty After Internal Fixation: A Machine-learning Algorithm. Clin Orthop Relat Res. 2022 Dec 1;480(12):2350-2360. doi: 10.1097/CORR.0000000000002283. Epub 2022 Jun 21. PMID 35767811
- [Derived] Fixation using Alternative Implants for the Treatment of Hip fractures (FAITH) Investigators. Fracture fixation in the operative management of hip fractures (FAITH): an international, multicentre, randomised controlled trial. Lancet. 2017 Apr 15;389(10078):1519-1527. doi: 10.1016/S0140-6736(17)30066-1. Epub 2017 Mar 3. PMID 28262269
- [Derived] FAITH Investigators. Fixation using alternative implants for the treatment of hip fractures (FAITH): design and rationale for a multi-centre randomized trial comparing sliding hip screws and cancellous screws on revision surgery rates and quality of life in the treatment of femoral neck fractures. BMC Musculoskelet Disord. 2014 Jun 26;15:219. doi: 10.1186/1471-2474-15-219. PMID 24965132
- [Derived] Zielinski SM, Viveiros H, Heetveld MJ, Swiontkowski MF, Bhandari M, Patka P, Van Lieshout EM; FAITH trial investigators. Central coordination as an alternative for local coordination in a multicenter randomized controlled trial: the FAITH trial experience. Trials. 2012 Jan 8;13:5. doi: 10.1186/1745-6215-13-5. PMID 22225733

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were consented and then randomized. Some subjects were enrolled but dropped prior to randomization. Or withdrew after being randomized so no data was collected
Period: Overall Study
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws
Started | 557 | 551
Completed | 542 | 537
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws | Total
Number analyzed (Participants) | 542 | 537 | 1079
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (12.0) | 72.0 (12.3) | 72.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 327 | 657
  Male | 212 | 210 | 422
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 211 | 209 | 420
  Canada | 111 | 109 | 220
  United Kingdom | 7 | 9 | 16
  Netherlands | 121 | 126 | 247
  Norway | 11 | 12 | 23
  Germany | 2 | 2 | 4
  India | 62 | 63 | 125
  Australia | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Revision Surgery
Description: Additional Surgery on the affected hip
Time Frame: Measured 2 years after original surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws
Number analyzed (Participants) | 542 | 537
Participants | 107 | 117

2. Secondary Outcome: Quality of Life
Description: The SF-12 PCS is the short form - 12 Health Survey Physical component summary - 0 is bad and 100 is good The WOMAC is Western Ontario and McMaster Universities Osteoarthritis Index 0 is good and 100 is bad The EQ-5D is EuroQol5D 1 is good and 5 is bad
Time Frame: Measured 2 years after original surgery
Population: secondary outcomes not given or completed to all subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws
Number analyzed (Participants) | 235 | 224
units on a scale
  SF-12 PCS: number analyzed (Participants) | 207 | 181
  SF-12 PCS | 41.6 (10.9) | 41.4 (11.8)
  WOMAC: number analyzed (Participants) | 205 | 183
  WOMAC | 40.97 (16.33) | 39.75 (17.09)
  EQ-5D: number analyzed (Participants) | 232 | 207
  EQ-5D | 0.79 (0.19) | 0.80 (0.19)
Statistical Analysis 1: Comparison: Single Sliding Hip Screw vs Multiple Cancellous Screws; Test type: Superiority; Cox Proportional Hazard = .83, 95% CI 2-sided [.63 to 1.09]

3. Secondary Outcome: Complications, Including Avascular Necrosis, Nonunion, and Infection
Time Frame: Measured 2 years after original surgery
Measure: Number; unit: participants
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws
Number analyzed (Participants) | 542 | 537
participants
  AVN | 50 | 28
  Nonunion | 33 | 33
  Infection | 10 | 9
Statistical Analysis 1: Comparison: Single Sliding Hip Screw vs Multiple Cancellous Screws; Test type: Superiority; p = 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Single Sliding Hip Screw | Multiple Cancellous Screws
All-Cause Mortality (participants affected / at risk) | 2/542 | 8/537
Serious Adverse Events (participants affected / at risk) | 115/542 | 104/537
Other Adverse Events (participants affected / at risk) | 55/542 | 45/537
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Sliding Hip Screw (N=542) | Multiple Cancellous Screws (N=537)
Abnormal Blood Complications (Blood and lymphatic system disorders) | 12 (13) | 7 (8)
Altered mental Status (General disorders) | 4 (5) | 6 (10)
Cancer (General disorders) | 5 (5) | 3 (3)
Cardiovascular (Cardiac disorders) | 19 (31) | 18 (22)
Death (General disorders) | 2 (2) | 8 (8)
Digestive Events (Gastrointestinal disorders) | 8 (8) | 8 (8)
Fall (General disorders) | 2 (2) | 2 (2)
Hernia (General disorders) | 0 (0) | 1 (1)
Infection/Sepsis (Infections and infestations) | 6 (6) | 5 (8)
Other (General disorders) | 20 (25) | 12 (14)
Other fractures (Musculoskeletal and connective tissue disorders) | 5 (10) | 9 (12)
Pain (General disorders) | 4 (6) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 16 (40) | 11 (20)
Renal Disease/Events (Renal and urinary disorders) | 5 (6) | 5 (5)
UTI (Renal and urinary disorders) | 7 (8) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Sliding Hip Screw (N=542) | Multiple Cancellous Screws (N=537)
Acute Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Avascular Necrosis (Cardiac disorders) | 44 (65) | 30 (39)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Cancer (General disorders) | 7 (7) | 10 (10)
Cardiovascular Event (Cardiac disorders) | 5 (5) | 13 (14)
Deep Brain Thrombosis (General disorders) | 4 (4) | 4 (4)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Metal Allergy (General disorders) | 1 (1) | 0 (0)
Other (General disorders) | 1 (1) | 0 (0)
Pnuemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prolonged Hospitalization (General disorders) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Sepsis (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Surgeons and patients were not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No